CLINICAL TRIAL: NCT00633126
Title: Pharmacokinetics of a Single Dose of Ceftaroline in Subjects 12 to 17 Years of Age Receiving Antibiotic Therapy
Brief Title: Pharmacokinetics of Ceftaroline in Subjects 12 to 17 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P903-15
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Infection
Keywords: PK; Pharmacokinetics
MeSH Terms: conditions — Infections | interventions — Ceftaroline; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): ceftaroline
  Interventions: Drug: ceftaroline

INTERVENTIONS:
Drug: ceftaroline — Single parenteral infusion at a dose of 8 mg/kg for subjects weighing less than 75 kg or at a dose of 600 mg for subjects weighing greater than or equal to 75 kg infused over 60 minutes.
  Other Names: ceftaroline for injection; ceftaroline fosamil

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of ceftaroline in pediatric subjects

DETAILED DESCRIPTION:
The purpose of this study is to determine the pharmacokinetics profile of ceftaroline in pediatric subjects

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized and receiving antibiotic therapy for treatment of a suspected infection of any type
* Body mass index (weight [kg]/height squared [m2]) of no more than 30
* Males and females between 12 and 17 years of age, inclusive

Exclusion Criteria:

* History of any hypersensitivity or allergic reaction to any β-lactam antimicrobial
* Past or current history of epilepsy or seizure disorder
* Critically ill or unstable patients

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Cerexa, Study Director — Forest Laboratories
Locations (4):
- United States (4):
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Durham, North Carolina
  - Investigational site, Akron, Ohio
  - Invetigational Site, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftaroline: Single group assignment, single dose of 600mg ceftaroline administered intravenously.
Period: Overall Study
Arm/Group | Ceftaroline
Started | 9
Completed | 8
Not Completed | 1
Not completed — Did not receive full dose | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ceftaroline
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.80)
Age, Customized [Number; unit: participants]
  <=18 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Plasma Concentration (Cmax) of Ceftaroline After Administration of Ceftaroline Fosamil at a Dose of 8 mg/kg up to a Maximum Dose of 600 mg Via IV Infusion Over 60 Minutes.
Description: The maximum plasma concentration (Cmax ) occurred around the time of the end of study drug infusion.
Time Frame: 12 hours after infusion
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ceftaroline
Number analyzed (Participants) | 8
ng/mL | 15276 (5997)

2. Secondary Outcome: Number of Adverse Events (AEs) Reported After Starting Study Drug Administration (Treatment Emergent Adverse Events, TEAEs) by Relationship to Ceftaroline (Related or Unrelated).
Description: A TEAE is any untoward medical occurrence a subject experiences following study drug administration.
  Subjects were monitored for TEAEs from the start of infusion of ceftaroline fosamil on Study Day 1 through the follow-up contact on Day 7.
Time Frame: Signing of Informed Consent Form (ICF) to last follow up (FU) visit, study day 7 (+-2 days).
Population: per protocol
  Out of 9 participants analyzed, 1 subject did not receive the full dose of study drug.
Measure: Number; unit: events
Arm/Group | Ceftaroline
Number analyzed (Participants) | 9
events | 8

ADVERSE EVENTS:
Time Frame: AEs were evaluated from the start of study drug infusion to last FU visit, study day 7 (+-2 days).
Description: Serious Adverse Events (SAEs) were evaluated through 30 days after the Ceftaroline infusion.
Arm/Group | Ceftaroline
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=9)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=9)
Vomiting (Gastrointestinal disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
ECG Prolonged QT (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No